CLINICAL TRIAL: NCT05353114
Title: Clinical Efficacy of a 3D Foot Scanner App for the Fitting of Therapeutic Footwear in Persons With Diabetes in Remission: A Randomized and Controlled Clinical Trial.
Brief Title: Clinical Efficacy of a 3D Foot Scanner for the Therapeutic Footwear Fitting
Acronym: Smartfitting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Jose Luis Lazaro Martinez, Prof. Dr, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CT-042022
Record Dates: First submitted 2022-04-22; First posted 2022-04-29 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Diabetic Foot; Orthopedic Disorder; Foot Ankle Injuries
Keywords: Prevention; Therapeutic footwear; New technologies
MeSH Terms: conditions — Diabetic Foot; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Therapeutic Footwear prescription group (No Intervention): 1) Patients that will acquire the therapeutic footwear size and model according to aesthetic preferences
- Therapeutic Footwear prescription based on a 3D Foot scanner (Experimental): 2) Patients that will acquire a specific size and model according to result of a novel mobile app 3D feet scan (smart-fitting by Podiapp - Podartis s.r.l Unipersonale-Crocceta del Montello (TV), Italy).
  Interventions: Other: 3D feet scan (smart-fitting by Podiapp - Podartis s.r.l Unipersonale-Crocceta del Montello (TV), Italy).

INTERVENTIONS:
Other: 3D feet scan (smart-fitting by Podiapp - Podartis s.r.l Unipersonale-Crocceta del Montello (TV), Italy). — The 3D foot scan becomes a movile app that recommends a specific size and model of therapeutic footwear according to the measurements
  Arms: Therapeutic Footwear prescription based on a 3D Foot scanner

SUMMARY:
Patients with diabetes at high risk of ulceration require a perfect fitting shoe to avoid high shear and pressure forces. Neuropathy skews sensory perceptions and can alter the proper selection of the therapeutic footwear.

The aims of study were to evaluate the ability of high-risk patients with diabetes in remission to select the proper therapeutic footwear and to validate a novel 3D foot scanner app for selecting the proper fitting therapeutic footwear.

DETAILED DESCRIPTION:
A Randomized Controlled Clinical Trial in 30 patients with a previous healed diabetic foot ulcer.

After parallel randomization (1:1) patients will be enrolled into two different groups:

1. Patients that will acquire the therapeutic footwear size and model according to aesthetic preferences;
2. Patients that will acquire a specific size and model according to result of a novel mobile app 3D feet scan (smart-fitting by Podiapp - Podartis s.r.l Unipersonale-Crocceta del Montello (TV), Italy).

Validation of proper therapeutic footwear fitting will be performed by a specialized podiatrist after acquisition of shoes in both groups.

Therapeutic Footwear will be recommended to change when following ill fitting reason been found: excessive length or tight, or compromise with toes

ELIGIBILITY:
Inclusion Criteria:

* High risk patients according to the International Working Group Diabetic Foot Guidelines (IWGDF-risk 3).
* Healed diabetic foot ulcer at the moment of inclusion.
* Capability to walk autonomously without walking aids.
* Diabetic Peripheral neuropathy.

Exclusion Criteria:

* Major amputation in the contralateral limb (below or above the knee).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure was the requirement of Therapeutic Footwear change after prescription because ill fitting. | 1 week
  Validation of proper therapeutic footwear fitting was performed by a specialized podiatrist after acquisition of shoes in both groups. TF was recommended to change when following ill fitting reason were found: excessive length or tight, or compromise with toes

SECONDARY OUTCOMES:
Number of participants with an ulcer occurrence event | 1 month
  Presence of a new o previous ulcer located in the foot in a patient with diabetes

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Universitaria de Podología de la Universidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No